CLINICAL TRIAL: NCT02847208
Title: Contraceptive Practices and Cervical Screening in Women With Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0489
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; contraception; gynaecological follow-up; screening; Pap smear; counselling
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cystic fibrosis women: It was a cohort of 155 CF women attending the Lyon adult centre. Women attending the CF adult centre in 2014 completed a written questionnaire about their contraceptive choices, frequency of gynaecological follow-up and cervical screening. Other clinical data were collected from the CF adult centre registry.
  Interventions: Other: self-report written questionnaire

INTERVENTIONS:
Other: self-report written questionnaire — The questionnaire was filled-in by the patients in presence of a clinical nurse. The gynaecological healthcare options and contraceptive choices were recorded. All following questions were closed-ended (answer yes/no): use of contraception; use of contraceptive pill; use of contraceptive implant; use of intrauterine device; use of tubal sterilization; use of mechanical contraception; use of other type of contraception; previous delivery (term pregnancy); gynaecological follow-up; previous Pap smear. In case of a positive answer to one of these questions, more details were requested (depending on the situation: name of the contraception, date of delivery, frequency of the gynaecological follow-up, date of the last pap smear). An internal validation of the questionnaire was performed on a subgroup of patients.

SUMMARY:
Little is known about gynaecological follow-up and cervical screening in Cystic Fibrosis (CF). Only few studies have described contraceptive practices in cohorts of CF women.

The investigators did a cross-sectional study in a cohort of 155 CF women attending the Lyon adult centre. Women attending the CF adult centre in 2014 completed a written questionnaire about their contraceptive choices, frequency of gynaecological follow-up and cervical screening. Other clinical data were collected from the CF adult centre registry.

One hundred and twenty women (100%) answered the questionnaire, among whom two were post-menopausal (46 and 59 years of age), and five were pregnant.

Seventy-four per cent of the women declared they had undergone gynaecological followup (89% of the women with transplantation), and only 55% reported having at least one previous Pap smear test. Among the transplanted patients, only 58% had had a Papsmear test, despite immunosuppressive treatment. The overall rate of contraception was only 64% and in diabetic women, it was 61%. Among contraception users; 65% used oral contraception, predominantly combined estrogen-progestagen (47%); among diabetic patients, 26% used progestin-only contraception. Intrauterine device accounted for 10% of patients using contraception, and tubal ligation only 4%.

This study is limited by its cross-sectional design. Despite an internal validation of the questionnaire showing an almost perfect agreement, the risk of recall bias has to be taken into account.

This study of practices highlights the importance of improved information regarding sexuality, fertility and reproductive health in young women with CF. A regular gynaecological follow-up and cervical screening is mandatory in this population.

Better gynaecological care and contraceptive advice would help to avoid unplanned pregnancies, and optimize contraceptive selection in relationship to specific clinical conditions.

ELIGIBILITY:
Inclusion Criteria:

* woman with cystic fibrosis
* followed in the Lyon adult centre in 2014

Exclusion Criteria:

- No exclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It was a cohort of 155 CF women attending the Lyon adult centre. Women attending the CF adult centre in 2014 completed a written questionnaire about their contraceptive choices, frequency of gynaecological follow-up and cervical screening. Other clinical data were collected from the CF adult centre registry.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a regular gynecological follow-up and cervical screening | At completion of the questionnaire (Day 1)

SECONDARY OUTCOMES:
Proportion of women using contraception and contraceptive type | At completion of the questionnaire (Day 1)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Rousset Jablonski, MD, Principal Investigator — Cystic Fibrosis Adult Referral Centre, Department of Internal Medicine, Centre Hospitalier Lyon Sud, Hospices Civils de Lyon
Locations (1):
- Cystic Fibrosis Adult Referral Centre, Department of Internal Medicine, Centre Hospitalier Lyon Sud, Hospices Civils de Lyon, Pierre-Bénite, France